CLINICAL TRIAL: NCT05356455
Title: The Effect of Motivational Interviewing Technique on Loneliness Levels in University Students Aged 18-25 Living Far From Home : Randomized Controlled Study
Brief Title: Motivational Interviewing Technique on Loneliness Levels in University Students Aged 18-25 Living Far From Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Aykut Karademir, Nurse, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KTO KaratayU - SBYH-01
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Loneliness
Keywords: Loneliness; Motivational interview technique; University students

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blind structures were sent to the statistician by grouping them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENT- active (Experimental): Motivational interview technique
  Interventions: Behavioral: motivational interview technique
- control passive (No Intervention): just watched

INTERVENTIONS:
Behavioral: motivational interview technique — Difference between pre-test and post-test
  Arms: EXPERIMENT- active

SUMMARY:
Purpose of the research This research was planned to evaluate the effect of motivational interview technique on loneliness in university students aged 18-25 living far from home.

DETAILED DESCRIPTION:
Loneliness is an unpleasant emotional state that needs to be investigated and examined, and can be perceived and defined in different ways in society. In addition, the most well-known definition of loneliness belongs to Peplau and Perlman (1984): According to Peplau and Perlman (1984), loneliness is an unpleasant feeling that causes anxiety and anxiety as a result of the inconsistency between the individual's existing social relationships and the social relationships he/she wishes to have or imagine. is the case. According to Weiss (1973), another important theorist, loneliness is the absence of desired social relationships or the absence of intimacy, intimacy and sensuality in these relationships despite having different social relationships.Loneliness is the deepest emotion and thought of the human mind. The only being who knows that he is alone, who is satisfied with this situation and even needs another person is human. Individuals who think of loneliness as a freedom and self-discovery can get lost in the depth of this feeling over time. While it may seem like a good way to generate solitude or recuperate your energy by taking time to listen to yourself, it is never completely healthy and effective. Because if the habitual loneliness becomes chronic, it can overwhelm the individual and make it destructive. The definition of this unpleasant emotional state and the way it is experienced in each person can be different. It is a virtuous and at the same time overwhelming emotional state. Loneliness actually gives very valuable information in getting to know people and interpreting life.

University years, which coincide with the late adolescence of 18-25 years, is a risky period with many problems such as staying away from home and family, adaptation to a new city, problems with education, uncertainties in becoming a candidate for a profession. The intensity of problems and expectations, the inadequacy of their families' social support prevent individuals from making correct assessments, lower their self-confidence and cause some mental problems. Anxiety, hopelessness and helplessness due to these problems push university students to loneliness. The young adult stage, called "developing adulthood", which ranges from 18 to 25 years of age, has higher risk-taking behavior, psychiatric disorders, and negative health behaviors than previous generations. Indeed, young adults' mental illness has increased in recent years, including anxiety and depression. In addition, many young adults have recently left their homes and families to attend university. Separation from their families has also prevented them from establishing long-term romantic relationships. As a result, levels of loneliness are high (up to 71% "sometimes" or "often" alone). In general, young adults struggle with a growing number of health problems. Many of these problems also occur during university years. Although most of the literature on loneliness focuses on older adults, many studies show that loneliness is especially common among younger generations. 43.3%, and 26% of university students stated that they would "never" or "rarely" find a friend when they needed it . As a result of this pushed loneliness, unwanted mental health problems such as depression and anxiety may occur.In recent years, interpersonal relations have deteriorated for some reasons and there has been a rapid increase in the number of people who lack intimacy and intimacy. Deterioration of interpersonal relations creates situations such as developing technology, fast lifestyles, frequent use of social media, virtual communication scattered with emojis and virtual dating . As a result of this, loneliness emerges as an important problem that negatively affects the life of the person and is increasing day by day. University students may experience loneliness due to being away from their families, and sometimes they may feel lonely even though they are with their friends. Therefore, the basis of loneliness can be the lack of social relationships and the inadequacy of satisfaction from these relationships. In addition, it is stated that university students in the young adult age group who experience the feeling of loneliness state less reasons to continue their lives, cause depression and anxiety, express a higher probability of suicide, and are more hopeless about the future. Therefore, when all these are taken into account, it has been seen that there is a meaningless and opposite relationship between the individual's attitudes towards protecting his own health and the feeling of loneliness. In addition, the increase in the perception of social support indirectly affects the sense of loneliness and public health by indirectly causing healthy behaviors. Contrary to the idea that loneliness will increase in later ages in the society and it is more common in the elderly, studies have shown that it is also common in young adults.Therefore, as there are university years between the ages of 18-25, it is seen that unpleasant feelings such as loneliness are experienced more frequently in this age range . Thinking about their future and their efforts to adapt to a new school, a new city and an unusual new environment for their dreams create different problems for many students, and these problems alienate university students from themselves. Considering all these situations , it is thought that it is an indispensable basic requirement for university students to take initiatives for university students to continue their social relations at the desired level, to eliminate the unpleasant feeling of loneliness they experience, to adapt to the environment and to maintain their psychological well-being.Looking at the results of the meta-analysis researched and attempted on loneliness, it is seen that the earliest study and research dates back to the 1930's. If we briefly talk about these researches and initiatives; It has been stated that it may be beneficial to develop social skills, increase social support, increase opportunities for social interaction, and address incompatible social cognition. When many studies are examined, when social skills are examined among university students who experience loneliness in general, the cause of loneliness is associated with self-consciousness and shyness. Finally, studies focusing on incompatible social cognition through Cognitive Behavioral Therapy have been found to be somewhat successful in reducing loneliness. It has been seen that the purpose of Cognitive Behavioral Therapy is to teach lonely individuals to identify negative thoughts, to associate them with reality and to distinguish them. When some studies are examined; Interventions focusing on social skills and social support showed promise for reducing loneliness. In fact, some studies have indicated that combining Cognitive Behavioral Therapy with social skills training is more effective in treating adults alone than treatment alone. All of the reviews noted the lack of randomized controlled trials and called for greater rigor in the evaluation of loneliness reduction interventions.It is thought that the Motivational Interview Technique on the loneliness experienced by university students who experience loneliness will be effective because it provides an initiative, an individual-oriented approach and awareness, similar to Cognitive Behavioral Therapy .

Motivational Interview Technique, which is an individual-centered and understanding oriented approach designed to motivate individuals who are not ready for change, provides its own internal motivation formation by solving the ambivalence of individuals towards changing behavior . In short, it is a technique that is used by making use of the individual's own internal motivation in order to realize the situation in which the person lives and to take action and action after being aware of it. When the randomized controlled studies with Motivational Interview Technique are examined, it is seen that it can be used in smoking, alcohol and substance use, drug use of chronic patients, post-traumatic conditions, diet compliance of Type 2 Diabetes patients, improving drug compliance of patients with hypertension, improving self-care in patients with depression and anxiety disorders and chronic heart failure. has been found to be effective meta-analyses are examined, it is stated that it is .Considering the meta-analyses, it was stated that it was effective even in very short interviews (15 minutes). Motivational Interview Technique is an approach that tries to understand the individual, as it questions the expectations, beliefs, future goals, and what he does for his goals. It is thought that it is very important for nurses, who work as the basic human power in health protection and development practices, to use Motivational Interview Technique, which is an individual-centered and effective approach, in nursing practices. For this reason, it is thought that Motivational Interview Technique will be effective in loneliness in order for individuals to be aware of their situation, to get rid of their ambivalent feelings and to take action to change. For this reason, it is considered important to conduct studies evaluating the effect of Motivational Interview Technique on loneliness and to test the effect of Motivational Interview Technique on loneliness.

ELIGIBILITY:
Inclusion Criteria:

Social and Emotional Loneliness Scale for Adults (Selsa-S) score above 45

* be between the ages of 18-25
* Living away from his family (home)
* KTO Karatay University Associate, undergraduate, graduate students

Exclusion Criteria:

* Knowing and applying motivational interviewing technique •Having a communication barrier for any reason (not knowing Turkish, etc.)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
The Effect of Motivational Interviewing Technique on Loneliness Levels in University Students aged 18-25 living far from home : Randomized Controlled Study | 2 weeks
  the result is not finished yet

CONTACTS AND LOCATIONS:
Overall Officials: Aykut Karademir, Nurse, Principal Investigator — Nurse
Locations (1):
- Aykut, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No